CLINICAL TRIAL: NCT03237741
Title: A Phase I Open-Label Study to Determine the Relative Bioavailability of GDC-0134 and to Investigate the Effect of Food and Proton Pump Inhibitor on Pharmacokinetics of GDC-0134 in Healthy Female Subjects of Non-childbearing Potential
Brief Title: Bioavailability of GDC-0134 and the Effect of Food and Proton Pump Inhibitor on Pharmacokinetics of GDC-0134 in Healthy Female Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: Quotient Clinical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GP39778; 2017-000299-27 (EudraCT Number)
Record Dates: First submitted 2017-07-31; First posted 2017-08-02 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Rabeprazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment Sequence 1: ABC1D1 (Experimental): Single dose of reference capsule GDC-0134 (Treatment A) during Period 1. Single dose of prototype capsule GDC-0134 (Treatment B) during Period 2. Single dose of GDC-0134 prototype capsule administered as GDC-0134-in-applesauce preparation under fasting conditions (Treatment C1) during Period 3. Single dose of GDC-0134 prototype capsule administered under fasting conditions in combination with 20 mg rabeprazole, and following prior administration of rabeprazole once daily for 3 days (Treatment D1) during Period 4. The washout period between doses will be a minimum of 21 days.
  Interventions: Drug: Reference capsule GDC-0134; Drug: Prototype capsule GDC-0134; Drug: rabeprazole
- Treatment Sequence 2: ABC2D2 (Experimental): Single dose of reference capsule GDC-0134 (Treatment A) during Period 1. Single dose of prototype capsule GDC-0134 (Treatment B) during Period 2. Single dose of GDC-0134 prototype capsule administered after a high-fat meal (Treatment C2) during Period 3. Single dose of GDC-0134 prototype capsule administered after a high-fat meal in combination with 20 mg rabeprazole, and following prior administration of rabeprazole once daily for 3 days (Treatment D2) during Period 4. The washout period between doses will be a minimum of 21 days.
  Interventions: Drug: Reference capsule GDC-0134; Drug: Prototype capsule GDC-0134; Drug: rabeprazole
- Treatment Sequence 3: BAC1D1 (Experimental): Single dose of prototype capsule GDC-0134 (Treatment B) during Period 1. Single dose of reference capsule GDC-0134 (Treatment A) during Period 2. Single dose of GDC-0134 prototype capsule administered as GDC-0134-in-applesauce preparation under fasting conditions (Treatment C1) during Period 3. Single dose of GDC-0134 prototype capsule administered under fasting conditions in combination with 20 mg rabeprazole, and following prior administration of rabeprazole once daily for 3 days (Treatment D1) during Period 4. The washout period between doses will be a minimum of 21 days.
  Interventions: Drug: Reference capsule GDC-0134; Drug: Prototype capsule GDC-0134; Drug: rabeprazole
- Treatment Sequence 4: BAC2D2 (Experimental): Single dose of prototype capsule GDC-0134 (Treatment B) during Period 1. Single dose of reference capsule GDC-0134 (Treatment A) during Period 2. Single dose of GDC-0134 prototype capsule administered after a high-fat meal (Treatment C2) during Period 3. Single dose of GDC-0134 prototype capsule administered after a high-fat meal in combination with 20 mg rabeprazole, and following prior administration of rabeprazole once daily for 3 days (Treatment D2) during Period 4. The washout period between doses will be a minimum of 21 days.
  Interventions: Drug: Reference capsule GDC-0134; Drug: Prototype capsule GDC-0134; Drug: rabeprazole

INTERVENTIONS:
Drug: Reference capsule GDC-0134 — Oral administration of a single dose of 200 milligrams (mg) GDC-0134 reference capsule administered as two 100 mg capsules.
Drug: Prototype capsule GDC-0134 — Oral administration of a single dose of 200 mg GDC-0134 prototype capsule administered as one 200 mg capsule.
Drug: rabeprazole — Oral administration of 20 mg rabeprazole once daily on Days -3, -2 and -1 as well as on Day 1 two hours prior to each administration of GDC-0134 during Period 4.

SUMMARY:
This study will evaluate the pharmacokinetics and safety of GDC-0134 in healthy female volunteers of non-childbearing potential. The first part of the study will compare the bioavailability of a prototype capsule of GDC-0134 relative to an existing GDC-0134 reference capsule (Periods 1 and 2). The second part of the study will assess the effect of GDC-0134-in-applesauce preparation under fasting conditions, the effect of low and high fat foods as well as the effect of elevated stomach pH via pre-treatment with rabeprazole, a proton pump inhibitor (PPI), under fasted and high-fat meal conditions (Periods 3 and 4).

ELIGIBILITY:
Inclusion Criteria:

* Healthy female participants between 30 and 65 years of age, inclusive;
* Within body mass index range 18.0 to 35.0 kilograms per square meter (kg/m^2), inclusive;
* Female participants will be of non-childbearing potential;
* In good health, determined by no clinically significant findings from medical history, 12-lead echocardiogram (ECG), and vital signs;
* Clinical laboratory evaluations within the reference range for the test laboratory, unless deemed not clinically significant by the investigator;
* Normal ophthalmology assessment.

Exclusion Criteria:

* Males and females of childbearing potential;
* Significant history or clinical manifestation of any significant metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal (GI), neurological, or psychiatric disorder (as determined by the investigator;
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the investigator;
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs;
* History of GI bleeding or GI ulcers;
* Any personal or family history of bleeding disorders, and any personal use of drugs known to affect blood clotting within 30 days of dosing;
* Any acute or chronic medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the subject's safe participation in and completion of the study.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2017-12-14 (Actual); Study Completion 2017-12-14 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve Extrapolated to Infinity (AUC0-inf) of GDC-0134 | Periods 1-4: Day 1: pre-dose, post-dose at 0.5 hours (h), 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h and 16 h, Day 2: post-dose 24 h and 36 h, Day 3, Day 4, Day 6, Day 8, Day 15 and Day 22
  The AUC0-inf is calculated in a plot of concentration of drug in blood plasma against time and extrapolated to infinity.
Area Under the Plasma Concentration-Time Curve up to Time Tau (AUC0-t) of GDC-0134 | Periods 1-4: Day 1: pre-dose, post-dose at 0.5 hours (h), 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h and 16 h, Day 2: post-dose 24 h and 36 h, Day 3, Day 4, Day 6, Day 8, Day 15 and Day 22
  The AUC0-t is calculated in a plot of concentration of drug in blood plasma against time and calculated up to the time of the last measurable GDC-0134 concentration.
Maximum Observed Concentration (Cmax) of GDC-0134 | Periods 1-4: Day 1: pre-dose, post-dose at 0.5 hours (h), 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h and 16 h, Day 2: post-dose 24 h and 36 h, Day 3, Day 4, Day 6, Day 8, Day 15 and Day 22
  Cmax is the maximum observed concentration of drug in blood plasma.
Time to Maximum Concentration (Tmax) of GDC-0134 | Periods 1-4: Day 1: pre-dose, post-dose at 0.5 hours (h), 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h and 16 h, Day 2: post-dose 24 h and 36 h, Day 3, Day 4, Day 6, Day 8, Day 15 and Day 22
  Tmax is the time elapsed from the time of drug administration to maximum plasma concentration.
Apparent Half-Life (t1/2) of GDC-0134 | Periods 1-4: Day 1: pre-dose, post-dose at 0.5 hours (h), 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h and 16 h, Day 2: post-dose 24 h and 36 h, Day 3, Day 4, Day 6, Day 8, Day 15 and Day 22
  Half-life is defined as the time required for the drug plasma concentration to be reduced to half.

SECONDARY OUTCOMES:
Percentage of Participants with Adverse Events | From baseline until 21 days after the last dose of study drug up to approximately 16 weeks
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Quotient Clinical Ltd, Clinical Research Unit, Nottingham, United Kingdom